CLINICAL TRIAL: NCT02653807
Title: The Immediate Effects of Two Manual Therapy Techniques on Ankle Musculoarticular Stiffness and Dorsiflexion Range of Motion in People With Chronic Ankle Rigidity: A Randomized Clinical Trial
Brief Title: Comparison of Two Manual Therapy Techniques on Ankle Dorsiflexion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Benjamin Hidalgo, visiting professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IREC/CARS-UCL-Hidalgo
Record Dates: First submitted 2016-01-05; First posted 2016-01-12 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Ankle Stiffness
Keywords: manual therapy; osteopathy; mobilization with movement; ankle; stiffness
MeSH Terms: interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mobilization with movement (Experimental): MWM at the talocrural joint during active weight bearing ankle dorsiflexion with the belt
  Interventions: Other: mobilization with movement
- osteopathic mobilization (Active Comparator): passive mobilization of the talo-crural joint
  Interventions: Other: osteopathic mobilization

INTERVENTIONS:
Other: mobilization with movement — manual therapy intervention
  Arms: mobilization with movement
Other: osteopathic mobilization — manual therapy intervention
  Arms: osteopathic mobilization

SUMMARY:
Ankle rigidity is a common musculoskeletal disorder affecting the talocrural joint, which can impair weight-bearing ankle dorsiflexion (WBADF). The objective was to compare the efficacy of Mulligan Mobilization with Movement (MWM) and Osteopathic Mobilization (OM) for improving ankle dorsiflexion range of motion (ROM) and musculoarticular stiffness (MAS).

DETAILED DESCRIPTION:
Increased musculoarticular stiffness (MAS) of the talocrural joint is a frequently encountered problem, identified during evaluation of weight bearing ankle dorsiflexion (WBADF). Such stiffness may follow ankle injury such as ankle sprain. In such a situation, MAS could be increased and might leads to a lack of joint flexibility as well as decreased dorsiflexion range-of-motion (ROM), however asymmetric rigidity does not necessarily always follow ankle sprain. Nevertheless, MAS is an important and necessary component of normal stability of the talocrural joint and could help to prevent abnormal ankle joint movement and ankle sprains.

Measurement of MAS can be determined by a technique known as free-oscillation, which is a comprehensive measure of joint stiffness comprising the stiffness of the muscle-tendon unit, skin, ligaments and joint capsule, along with a number of other mechanical and neuromuscular factors. The assessment of MAS is important when evaluating muscular performance, injury prevention and gender differences in flexibility. For example, men, as well as older people, are known to present with greater MAS than women and young people.

MAS of the talocrural joint can be objectively measured using an electromechanical device that imparts a passive oscillatory dorsiflexion movement, but also by means of clinical tests such as toe-wall distance and angular goniometric measurement during the weight bearing lunge test. Electromechanical measurement of ankle MAS has been used in several previous studies of asymptomatic participants and in patients with fibromyalgia syndrome, and spasticity after a stroke.

In orthopaedic manual therapy, different methods have been proposed to treat MAS associated with loss of dorsiflexion ROM at the talocrural joint. These include single session of Mulligan's Mobilization with Movement (MWM), anteroposterior mobilization of the talus, high velocity thrust, and Osteopathic Mobilization (OM). These methods have been described in clinical practice manuals, with greater proportion of studies reporting on the effects of MWM in comparison to high velocity thrust for improving ankle dorsiflexion ROM in chronic ankle instability or to study MWM efficacy in isolation for subacute or recurrent ankle sprains and for chronic ankle instability. With the exception of one study the results are generally in favor of MWM.

Generally MWM is an increasingly popular form of manual therapy for musculoskeletal disorders, concerning the ankle MWM try to improve talocrural ROM. MWM is a combination of accessory joint glide of the talus combined with active ankle dorsiflexion movement. The patient performs active WBADF while the therapist simultaneously applies an anteroposterior glide of the talus with respective posteroanterior tibial glide with the aid of a manual therapy belt. OM is a purely passive anteroposterior mobilization of the talus with respect to tibia, performed in a non weight-bearing position. To date, there have been no studies comparing the effectiveness of each technique with respect to electromechanically determined ankle MAS or ankle joint ROM determined by the WBADF lunge test.

Therefore, the aim of the study was to investigate the relative efficacy of MWM and OM on MAS as the primary outcome measurement and joint ROM during the WBADF lunge test as the secondary outcome measurement. The hypothesis was that MWM would produce significantly greater reduction in MAS and increased ankle joint ROM when compared to OM.

ELIGIBILITY:
Inclusion Criteria:

* male gender, aged between 18 to 40 years, with a chronic unilateral mobility deficit of the talocrural joint; i.e. subjective blocking sensation and/or feeling of ankle stiffness together with the presence of ankle region pain/tenderness, during active WBADF while squatting. Subjects were recruited with chronic unilateral mobility deficit of the talocrural joint, which could be following a previous history of ankle injury or without previous history of ankle injury.

Exclusion Criteria:

* a history of ankle joint surgery or injury to the foot, ankle, knee or hip in the previous one-year.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Electromechanical device measurement of MAS (Lehmann device, 1989) | Change from baseline until discharge of treatment (same day, single session)
  The electromechanical device used to quantify musculoarticular stiffness had been used in previous research studies and has ben shown to have high precision, reliability and accuracy. An oscillating footplate produces passive ankle joint dorsiflexion with 5° amplitude sinusoidal rotary displacements. Thirty trials of 10 different oscillation frequencies, varying from 3 to 12 Hz, were applied on each subject during each session. See Detrembleur and Plaghki (2000) for more details of the process.

SECONDARY OUTCOMES:
WBAD lunge test | Change from baseline until discharge of treatment (same day, single session)
  the weight bearing ankle dorsiflexion lunge test a common clinical test used to evaluate ankle dorsiflexion ROM (Powden et al., 2015) which has been shown to have moderate to excellent intra-rater reliability (ICC = 0,65-0,99) with a minimal detectable change of 1,9 cm and 4,7°. A graduated tape measure was placed on the floor, perpendicular to the wall. The investigator demonstrated the measurement procedure test to the subject providing standardized instructions. The subject placed his symptomatic foot with the big toe aligned on the tape measure and performed ankle dorsiflexion until his knee touched the wall. An iPhone was used to measure the degree of tibial inclination.

CONTACTS AND LOCATIONS:
Locations (1):
- IREC/CARS - Tour Pasteur - Saint-Luc Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleyenheuft C, Detrembleur C, Deltombe T, Fomekong E, Lejeune TM. Quantitative assessment of anaesthetic nerve block and neurotomy in spastic equinus foot: a review of two cases. J Rehabil Med. 2008 Nov;40(10):879-81. doi: 10.2340/16501977-0263. PMID 19242629
- [Background] Dierick F, Detrembleur C, Trintignac G, Masquelier E. Nature of passive musculoarticular stiffness increase of ankle in female subjects with fibromyalgia syndrome. Eur J Appl Physiol. 2011 Sep;111(9):2163-71. doi: 10.1007/s00421-011-1850-2. Epub 2011 Feb 6. PMID 21298443
- [Background] Gilbreath JP, Gaven SL, Van Lunen L, Hoch MC. The effects of mobilization with movement on dorsiflexion range of motion, dynamic balance, and self-reported function in individuals with chronic ankle instability. Man Ther. 2014 Apr;19(2):152-7. doi: 10.1016/j.math.2013.10.001. PMID 24834500
- [Background] Hidalgo B, Pitance L, Hall T, Detrembleur C, Nielens H. Short-term effects of Mulligan mobilization with movement on pain, disability, and kinematic spinal movements in patients with nonspecific low back pain: a randomized placebo-controlled trial. J Manipulative Physiol Ther. 2015 Jul-Aug;38(6):365-74. doi: 10.1016/j.jmpt.2015.06.013. Epub 2015 Jul 26. PMID 26215900
- [Background] Lehmann JF, Price R, deLateur BJ, Hinderer S, Traynor C. Spasticity: quantitative measurements as a basis for assessing effectiveness of therapeutic intervention. Arch Phys Med Rehabil. 1989 Jan;70(1):6-15. PMID 2916921
- [Background] Marron-Gomez D, Rodriguez-Fernandez AL, Martin-Urrialde JA. The effect of two mobilization techniques on dorsiflexion in people with chronic ankle instability. Phys Ther Sport. 2015 Feb;16(1):10-5. doi: 10.1016/j.ptsp.2014.02.001. Epub 2014 Feb 14. PMID 24679362
- [Background] Powden CJ, Hoch JM, Hoch MC. Reliability and minimal detectable change of the weight-bearing lunge test: A systematic review. Man Ther. 2015 Aug;20(4):524-32. doi: 10.1016/j.math.2015.01.004. Epub 2015 Jan 29. PMID 25704110
- [Background] Suydam SM, Soulas EM, Elliott DM, Silbernagel KG, Buchanan TS, Cortes DH. Viscoelastic properties of healthy achilles tendon are independent of isometric plantar flexion strength and cross-sectional area. J Orthop Res. 2015 Jun;33(6):926-31. doi: 10.1002/jor.22878. Epub 2015 Apr 27. PMID 25882209
- [Background] Vicenzino B, Branjerdporn M, Teys P, Jordan K. Initial changes in posterior talar glide and dorsiflexion of the ankle after mobilization with movement in individuals with recurrent ankle sprain. J Orthop Sports Phys Ther. 2006 Jul;36(7):464-71. doi: 10.2519/jospt.2006.2265. PMID 16881463
- [Background] Ditroilo M, Watsford M, Murphy A, De Vito G. Assessing musculo-articular stiffness using free oscillations: theory, measurement and analysis. Sports Med. 2011 Dec 1;41(12):1019-32. doi: 10.2165/11591470-000000000-00000. PMID 22060176
- [Background] Collins N, Teys P, Vicenzino B. The initial effects of a Mulligan's mobilization with movement technique on dorsiflexion and pain in subacute ankle sprains. Man Ther. 2004 May;9(2):77-82. doi: 10.1016/S1356-689X(03)00101-2. PMID 15040966
- [Background] Teixeira LM, Pires T, Silva RD, de Resende MA. Immediate effect of a single anteroposterior talus mobilization on dorsiflexion range of motion in participants with orthopedic dysfunction of the ankle and foot. J Manipulative Physiol Ther. 2013 Jul-Aug;36(6):369-75. doi: 10.1016/j.jmpt.2013.06.003. Epub 2013 Jul 11. PMID 23850371
- [Background] Cejudo A, Sainz de Baranda P, Ayala F, Santonja F. A simplified version of the weight-bearing ankle lunge test: description and test-retest reliability. Man Ther. 2014 Aug;19(4):355-9. doi: 10.1016/j.math.2014.03.008. Epub 2014 Apr 2. PMID 24746162
- [Background] Bennell KL, Talbot RC, Wajswelner H, Techovanich W, Kelly DH, Hall AJ. Intra-rater and inter-rater reliability of a weight-bearing lunge measure of ankle dorsiflexion. Aust J Physiother. 1998;44(3):175-180. doi: 10.1016/s0004-9514(14)60377-9. PMID 11676731